CLINICAL TRIAL: NCT03330613
Title: Emergence Delirium and Recovery Time in Children: a Randomized Trial to Compare Total Intravenous Anesthesia With Propofol to Inhalational Sevoflurane Anesthesia for Ambulatory Dental Surgery
Brief Title: Emergence Delirium and Recovery Time in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ozlem Kocaturk, Asist.Prof. MD, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2017/17
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhalational anesthesia (Other): Inhalational anesthesia is an anesthesia procedure using by respiratory tract. PAEDS used to for postanesthesia pediatric patients.
  Interventions: Diagnostic Test: PAEDS; Procedure: TIVA; Procedure: Inhalational anesthesia
- Total intravenous anesthesia (Active Comparator): Total intravenous anesthesia (TIVA) is an anesthesia procedure using vascular infusion method.PAEDS used to for postanesthesia pediatric patients.
  Interventions: Diagnostic Test: PAEDS; Procedure: TIVA; Procedure: Inhalational anesthesia

INTERVENTIONS:
Diagnostic Test: PAEDS — pediatric emergency delirium scale
Procedure: TIVA — Total intravenous anesthesia with propofol
Procedure: Inhalational anesthesia — Inhalational (volatile) anesthesia with sevoflurane

SUMMARY:
In this study, inhalation anesthesia procedure and intravenous anesthesia method will be compared in terms of emergence delirium and recovery time in children who are scheduled for dental treatment under general anesthesia.

DETAILED DESCRIPTION:
Pediatric Anesthesia Early Delirium Scale (PAEDS) will be used to evaluate postoperative emergence delirium.

ELIGIBILITY:
Inclusion Criteria:

1. Indication of dental treatment under general anesthesia.
2. No systemic disease (ASA1).
3. Child and parent agree to participate in the work

Exclusion Criteria:

1. Do not accept to participate in the work.
2. The child is not systemically healthy.
3. Children with allergies to general anesthetic drugs.
4. Contraindicated children to take general anesthesia
5. Children with upper respiratory tract infection on the day of operation

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-07-15 (Estimated); Study Completion 2018-07-20 (Estimated)

PRIMARY OUTCOMES:
Emergence delirium | 6 hours
  Pediatric Anesthesia Early Delirium Scale (PAED) will be used to assess postoperative agitation.
  Point Description Not at all Just a little Quite a bit Very much Extremely
  1. The child makes eye contact with the caregiver 4 3 2 1 0
  2. The child's actions are purposeful 4 3 2 1 0
  3. The child is aware of his/her surroundings 4 3 2 1 0
  4. The child is restless 0 1 2 3 4
  5. The child is inconsolable 0 1 2 3 4
  The Pediatric Anesthesia Emergence Delirium Scale

SECONDARY OUTCOMES:
Recovery time | 6 hours
  The period of stay at the post-anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Kocaturk, Principal Investigator — Faculty of Dentistry, Adnan Menderes University
Locations (1):
- Ozlem Kocaturk, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandler JR, Myers D, Mehta D, Whyte E, Groberman MK, Montgomery CJ, Ansermino JM. Emergence delirium in children: a randomized trial to compare total intravenous anesthesia with propofol and remifentanil to inhalational sevoflurane anesthesia. Paediatr Anaesth. 2013 Apr;23(4):309-15. doi: 10.1111/pan.12090. PMID 23464658
- [Background] Konig MW, Varughese AM, Brennen KA, Barclay S, Shackleford TM, Samuels PJ, Gorman K, Ellis J, Wang Y, Nick TG. Quality of recovery from two types of general anesthesia for ambulatory dental surgery in children: a double-blind, randomized trial. Paediatr Anaesth. 2009 Aug;19(8):748-55. doi: 10.1111/j.1460-9592.2009.03054.x. Epub 2009 Jun 15. PMID 19538532